CLINICAL TRIAL: NCT03564600
Title: Optimizing Outcomes for Older Veterans With Chronic Low Back Pain Syndrome: Aging Back Clinics
Brief Title: Aging Back Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: O2808-R
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Chronic Low Back Pain
Keywords: low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABC Group (Experimental): Veterans with back pain for at least the past 6 months receive personalized care by providers trained based on a published set of algorithms that guide care for conditions that contribute to disability in older adults with chronic low back pain
  Interventions: Other: Aging Back Clinics management
- UC Group (No Intervention): Veterans with back pain for at least the past 6 months who receive usual care as directed by their primary care physician.

INTERVENTIONS:
Other: Aging Back Clinics management — Personalized care is delivered that is guided by published algorithms for each component condition identified by a trained provider.
  Arms: ABC Group

SUMMARY:
The purpose of this study is to compare two different ways to treat chronic low back pain. The two types of treatment that the investigators will compare are called Usual Care and ABC Care. Usual Care tends to focus on the spine. ABC Care focuses on the entire body and the mind. With Usual Care, participants will work with their own doctor to come up with a treatment plan. With ABC Care, participants will work with the investigators' ABC providers and their team. The investigators believe ABC Care will help reduce pain, lower costs, and increase participants' ability to do the things they enjoy doing better than Usual Care. In ABC Care the investigators hope to avoid treatments like surgeries where participants get metal rods put in their back.

This research is being done at three Veterans Hospitals: the Veterans Administration of Pittsburgh Healthcare System (VAPHS) in Pittsburgh, PA; the North Texas VA Medical Center in Dallas, TX; and the Hunter Holmes McGuire VA Medical Center in Richmond, VA. This research study is being paid for by the Rehabilitation Research and Development section of the Veterans Health Administration.

The investigators will be enrolling about 450 participants at 3 sites or around 150 at each site.

DETAILED DESCRIPTION:
Degenerative disease of the lumbar spine is ubiquitous in older adults, but low back pain is not. Treatments that focus exclusively on degenerative spine disease, such as spinal injection and surgery, have resulted in rising costs and exposure to potentially life-threatening morbidity but outcomes have not improved. The investigators posit that to improve treatment outcomes for older adults with chronic low back pain (CLBP - back pain that has been present on at least half the days for at least 6 months), the condition should be approached as a syndrome, that is, a final common pathway for the expression of many contributors, in the same way that geriatricians approach the evaluation and treatment of delirium and falls. Using this model, the lumbar spine is considered a weak link, but is rarely the sole treatment target. Conditions that commonly contribute to pain and disability in older adults with CLBP include hip osteoarthritis, fibromyalgia, anxiety, maladaptive coping, and myofascial pain, each of which is associated with specific evidence-based treatments. Because such conditions are not routinely evaluated in patients with CLBP, it is perhaps not surprising that first line treatments that do not specifically target multiple contributors (e.g. spine-focused physical therapy and analgesics) often provide suboptimal treatment outcomes. This often results in continued treatment-seeking including potentially toxic medications and invasive, expensive, and potentially life-threatening procedures such as complex spinal fusion.

The central question that the proposed randomized trial is designed to answer is: What is the efficacy of caring for older adults with CLBP in Aging Back Clinics (ABC), where the patient is first treated as an older adult, and second as a patient with CLBP, compared with usual care (UC)? The investigators have developed evidence and expert-opinion based guidelines for the evaluation and treatment of 12 key contributors to pain and disability in older adults with CLBP. The investigators' prior work also supports the commonplace nature of multiple contributors to CLBP in older Veterans and the feasibility of delivering patient-centered comprehensive care that follows the investigators' published guidelines. The investigators now wish to implement these guidelines in the investigators' ABC clinics and compare this approach to that of UC in older Veterans. Proof of the hypotheses could significantly impact patient care by reducing pain and disability and identifying key conditions whose treatment could prevent the pursuit of invasive treatments and their associated potential morbidity and cost.

About 450 Veterans age 65-89 with CLBP will be recruited from primary care provider practices at 3 VAs - VA Pittsburgh Healthcare System, Dallas VA, and Richmond VA to meet a target randomization of 330. Individuals will be randomized to receive either ABC care or UC and they will be followed for one year. Those in ABC care will be referred to a generalist (e.g., geriatrician, physiatrist, rheumatologist) that has been identified and trained in a structured assessment to identify the conditions for which evidence and expert opinion-based algorithms have been created. Usual care will not be constrained. Outcomes will be assessed at baseline and over the telephone at three later time points: 6 months, 9 months and 12 months. Health Care Utilization will be assessed monthly. Gait speed, a strong predictor of morbidity and mortality in older adults, will be measured at baseline. The proposed clinical trial has the potential not only to improve pain-related disability, but also to reduce morbidity, increase quality of life, and limit healthcare utilization.

ELIGIBILITY:
Inclusion Criteria:

* Older Veterans with CLBP, defined as pain in the lower back of at least moderate severity.

  * assessed with a verbal rating scale on > half the days for > 6 months
* Veterans must be English speaking.
* Must be able to commit to 12 months of study participation.
* The Quick Mild Cognitive Impairment Screen (QMCI) will be administered on site to screen for mild cognitive impairment (MCI).

  * Those with MCI will not be excluded, but their PCP will be alerted.

Exclusion Criteria:

* Positive screen for dementia (score <23 on the MMSE)
* Pain in other body locations that is more severe than their low back pain
* Red flags indicative of serious underlying illness requiring urgent care

  * e.g., fever, change in bowel/bladder function, sudden severe change in pain, unintentional weight loss, new lower extremity weakness
* Previous lumbar surgery.
* Acute illness.
* Psychotic symptoms.
* Prohibitive communication impairment.

  * e.g., severe hearing or visual impairment.
* Neither pregnant subjects nor women of childbearing potential will be included due to the age requirements of the study.
* Vulnerable subjects will not be enrolled, nor children and prisoners.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 299 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra K. Weiner, MD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (3):
- United States (3):
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABC Group | UC Group
Started | 150 | 149
Completed | 113 | 99
Not Completed | 37 | 50

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABC Group | UC Group | Total
Number analyzed (Participants) | 150 | 149 | 299
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 150 | 149 | 299
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (5.1) | 73.3 (5.0) | 73.39 (5.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 20
  Male | 136 | 143 | 279
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 14 | 25
  Not Hispanic or Latino | 139 | 135 | 274
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 41 | 41 | 82
  White | 105 | 99 | 204
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 150 | 149 | 299
Oswestry Disability Index [Mean (Standard Deviation); unit: units on a scale] — Range 0 to 100 with higher score indicating greater disability.
  units on a scale | 30.5 (14.7) | 33.1 (15.3) | 31.8 (15.02)

OUTCOME MEASURES:

1. Primary Outcome: Oswestry Disability Index (ODI) Change
Description: The ODI assesses interference of pain with function. This questionnaire is used by clinicians and researchers to quantify disability for low back pain. Range 0 to 100 with higher score indicating greater disability.
Time Frame: Baseline visit, every three months for up to one year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABC Group | UC Group
Number analyzed (Participants) | 150 | 149
units on a scale
  3 months | -0.4 (13.0) | 2.7 (11.3)
  6 months | -0.8 (12.0) | 1.2 (11.5)
  9 months | 1.3 (14.7) | -0.2 (12.6)
  12 months | 0.2 (14.0) | 2.8 (12.1)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | ABC Group | UC Group
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/149
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/149
Other Adverse Events (participants affected / at risk) | 0/150 | 0/149

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT03564600/Prot_SAP_000.pdf